CLINICAL TRIAL: NCT05974280
Title: Pilot Study on the Treatment of Anal Fistulas in Crohn's Disease Patients Using Alofisel Versus Fat Autologous Stem Cells
Brief Title: Study on the Treatment of Anal Fistulas Using Alofisel Versus Fat Autologous Stem Cells
Acronym: CHAZAM
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_CHAzAM_ED_001
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease; Anal Fistula
MeSH Terms: conditions — Crohn Disease; Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alofisel group (routine care): The patient receives Alofisel injection as in routine care
  Interventions: Drug: Alofisel
- Autologous fat injection (routine care): The back-up patient receives autologous fat stem cells injection as in routine care
  Interventions: Drug: Fat stem cell

INTERVENTIONS:
Drug: Alofisel — Alofisel is made up of 'mesenchymal stem cells' from the fat tissue of a donor. Alofisel is a medicine that is used to treat complex anal fistulas in adults with Crohn's disease
  Other Names: mesenchymal stem cells
  Groups: Alofisel group (routine care)
Drug: Fat stem cell — mesenchymal stem cells from adipose (fat) tissue injection
  Other Names: Fat graft
  Groups: Autologous fat injection (routine care)

SUMMARY:
One of the newest and most innovative medicinal approaches is cell therapy. Several clinical trials and experimental investigations have looked into the feasibility of treating CD-related fistulas with stem cells.

The current indication for ALOFISEL® (active ingredient: Darvadstrocel) is the treatment of difficult perianal Crohn's fistulas that have not responded well to at least one conventional therapy or biotherapy.

This brand-new cell therapy medication is created using amplified allogeneic human adult mesenchymal stem cells from adipose tissue (ADSC). The supplier mandates that two patients be booked for a single dose of ALOFISEL® due to the medication's expensive price-roughly €54,000 for a single dose of 120 million-which cannot be stored once thawed.

Only one of the two patients receives therapy; the other serves as the backup patient. By doing this, another "back-up" patient who might receive no care at all is avoided.

An developing alternate approach to allogeneic ADSC injection for the treatment of complicated anal fistulas in CD is autologous fat injection. In recent years, autologous fat grafts have been the subject of in-depth research. They are popular because it is simple to get clinical samples (lipoaspirate, adipose tissue), and because there are a lot of ADSCs in adipose tissue. Additionally, ADSCs show strong immunomodulatory and regenerative capacities.

We would wish to compare the effectiveness of these two injection kinds on perianal fistulas as part of our care of CD.

DETAILED DESCRIPTION:
The trial will be made available to patients who are scheduled for perianal surgery with ALOFISEL® or backup (fat injection). The history and signs of perianal fistula will be noted if the patient doesn't object.

Two visits that correspond to typical follow-up visits for patients will be noted:

Visit following surgery: fistula clinical evaluation, analgesic use, etc. and six months after : clinical assessment, MRI

ELIGIBILITY:
Inclusion Criteria:

* Complex anal fistula with the following criteria: - Inactive/slightly active luminal Crohn's disease under conventional treatment or biotherapy MRI has demonstrated effective drainage. Maximum of two internal orifices and three external orifices; persists despite internal orifice(s) closing.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients hypersensitive to the product, bovine serum or any of the excipients of Alofisel
* Vulnerable persons: deprived of liberty, under guardianship, under curatorship, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with Crohn's disease coming to the digestive surgery department of the CHU in Nantes for perianal surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparing the efficacy of Alofisel treatment versus fat grafting in Crohn's disease complex perianal fistulae | 1 month after the surgery
  At 1 month, the percentage of healing is defined as the clinical closure of the orifice and the lack of pus draining by pressure on the borders of the fistula scar.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France